CLINICAL TRIAL: NCT06013137
Title: Testing an Artificial Intelligence Chatbot for Mental Health
Brief Title: Chatbot for Depression, Anxiety, and Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Nicholas C. Jacobson, Dr. Nicholas Jacobson, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY02000591
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Depression; Anxiety; Eating Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): This group will have access to the Therabot smartphone application. They will interact with the generative chatbot daily to discuss their mental health. Each participant in this group will have some benchmark symptoms of depression, anxiety, or eating disorders. They will fill out questionnaires every 4 weeks to describe changes in symptoms.
  Interventions: Other: Therabot
- Control (No Intervention): This group will not have access to the Therabot App. They will fill out questionnaires every 4 weeks to describe changes in symptoms. Each participant in this group will have some benchmark symptoms of depression, anxiety, or eating disorders.

INTERVENTIONS:
Other: Therabot — The participants assigned to the experimental group will interact with an artificial intelligence therapy chatbot to alleviate symptoms associated with depression, anxiety, and eating disorders. The control group will not have access to this smartphone chatbot app.
  Other Names: Artificial Intelligence Chatbot
  Arms: Experimental

SUMMARY:
The research team would like to test how efficacious an artificial intelligence chatbot is in delivering supportive behavioral interventions in populations with anxiety, depression, or eating concerns.

DETAILED DESCRIPTION:
The research team has developed a deep learning-powered application that can provide support and therapeutic suggestions via natural dialogue. The chatbot is designed to be highly scalable such that it could address access issues (to address the majority of persons who do not not have access to therapy). Eventually, it is hoped this intervention can provide accessible therapy for those with anxiety, depression, and eating disorders, among other mental illnesses. The chatbot has been trained with intervention-oriented text conversations written by research assistants, employing a variety of therapeutic techniques, including cognitive-behavioral therapy. The research team hopes to test how well the chatbot can respond and aid those with mental health symptoms. The chatbot's effectiveness will be monitored based on the participants' interactions with the chatbot, as well as the participants' scores on the PHQ-9, GAD-IV, SWED, and general satisfactory questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit participants online using Facebook, Google Ads, Reddit, MTurk, listservs, and other online platforms.
* These individuals must meet the criteria for anxiety, depression or disordered eating, according to the PHQ-9, GADQ-IV, and SWED 3.0.

Exclusion Criteria:

* Individuals currently being treated for active suicidality (measured with C-SSRS), Bipolar I/II, and active psychosis will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Anxiety Symptoms | Each participant in the anxiety cohort will fill out an anxiety questionnaire to establish baseline symptoms, and they will fill out this questionnaire again after 4 and 8 weeks of using the therapy chatbot to track changes in their symptoms.
  Anxiety symptoms will be measured with the GAD-IV.
Depressive Symptoms | Each participant in the depression cohort will fill out a questionnaire to establish baseline symptoms, and they will fill out this questionnaire again after 4 and 8 weeks of using the therapy chatbot to track changes in their symptoms.
  Depressive symptoms will be measured with the PHQ-9.
Eating Disorders Symptoms | Each participant in the eating disorders cohort will fill out a questionnaire to establish baseline symptoms, and they will fill out this questionnaire again after 4 and 8 weeks of using the therapy chatbot to track changes in their symptoms.
  Eating Disorders symptoms will be measured with the SWED.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Jacobson, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth College, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No